CLINICAL TRIAL: NCT01940614
Title: Use of Copeptin in the Differential Diagnosis of Diabetes insipidus-a Prospective International Study
Brief Title: Use of Copeptin in Diabetes Insipidus
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: CODDI2013
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Diabetes Insipidus; Primary Polydipsia
Keywords: Copeptin; differential diagnosis of polyuria polydipsia syndrome; diabetes insipidus; compulsive water drinking; water deprivation test; Diabetes insipidus (central and nephrogenic)
MeSH Terms: conditions — Diabetes Insipidus; Polydipsia, Psychogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Water deprivation test — Classical water deprivation test alone
Other: Water deprivation test — classical water deprivation test plus plasma copeptin cut-off levels
Other: Hypertonic saline infusion — hypertonic saline infusion test plus plasma copeptin measurement

SUMMARY:
Prospective evaluation of the novel biomarker copeptin in the differential diagnosis of diabetes insipidus against the standard diagnostic test methods.

DETAILED DESCRIPTION:
Purpose of this study is to compare the overall diagnostic accuracy of the three following diagnostic test procedures in diabetes insipidus (central, nephrogenic) and primary polydipsia: a) classical water deprivation test alone, b) classical water deprivation test plus plasma copeptin cut-off levels, c) hypertonic saline infusion test plus plasma copeptin measurement.

The investigators hypothesize that firstly b) and c) is better as a). Secondly the investigators hypothesize that c) is non-inferior to b).

ELIGIBILITY:
Inclusion Criteria:

* Polyuria or/and Polydipsia or/and therapy with synthetic adenovirus proteinase (AVP) derivate
* Urine osmolality <800mOsm/kgH20

Exclusion Criteria:

* Polyuria due to diabetes mellitus
* Hypokalemia
* Hyperkalemia (>5mmol/l)
* Hypercalcemia
* Kidney disease (min.: glomerular filtration rate (GFR) 60ml/min/1.73m2)
* Pregnancy
* Hyponatremia >135mmol/L
* Hypernatremia >145mmol/L
* Hypo- or hypervolemia
* uncorrected adrenal or thyroidal deficiency
* Cardia failure
* Epilepsia
* Uncontrolled hypertension

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care center
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overall diagnostic accuracy | beginning and end of protocol, up to 9hours
  Ratio of the number of correctly diagnosed patients to the number of all tested patients for the tests:
  * classical water deprivation test alone
  * classical water deprivation test plus plasma copeptin cut-off levels
  * hypertonic saline Infusion test plus plasma copeptin measurements

SECONDARY OUTCOMES:
Sensitivity, specificity, positive and negative predictive value | beginning and end of protocol, up to 9hours
  each diagnostic test
post-hoc best copeptin cut-off optimising overall performance | beginning and end of protocol, up to 9hours
  best copeptin cut-offs for differentiation between different diagnosis of polyuria-polydipsia syndrome
subjective burden as rated by patients on visual analogue scale | beginning, during and end of protocol, up to 9hours
  water deprivation test and hypertonic saline Infusion test
Predictive value of specific anamnestic and clinical features | before tests
  Evaluation of anamnestic and clinical features to test-independently predict final diagnosis of polyuria-polydipsia syndrome
Predictive value of absent bright spot in posterior pituitary enlargement | before or after tests
  Evaluation of predictive value of absent bright spot in T1 weighted cranial MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Principal Investigator — University Hospital
Locations (1):
- Univerisity Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Atila C, Chifu I, Drummond JB, Vogt DR, Nahum U, Fassnacht M, Winzeler B, Refardt J, Christ-Crain M. A novel diagnostic score for diagnosing arginine vasopressin deficiency (central diabetes insipidus) or primary polydipsia with basal laboratory and clinical parameters: results from two international multicentre prospective diagnostic studies. Lancet Diabetes Endocrinol. 2025 Jun;13(6):505-515. doi: 10.1016/S2213-8587(25)00053-1. Epub 2025 Apr 25. PMID 40294614
- [Derived] Sailer CO, Refardt J, Blum CA, Schnyder I, Molina-Tijeras JA, Fenske W, Christ-Crain M. Validity of different copeptin assays in the differential diagnosis of the polyuria-polydipsia syndrome. Sci Rep. 2021 May 12;11(1):10104. doi: 10.1038/s41598-021-89505-9. PMID 33980941
- [Derived] Fenske W, Refardt J, Chifu I, Schnyder I, Winzeler B, Drummond J, Ribeiro-Oliveira A Jr, Drescher T, Bilz S, Vogt DR, Malzahn U, Kroiss M, Christ E, Henzen C, Fischli S, Tonjes A, Mueller B, Schopohl J, Flitsch J, Brabant G, Fassnacht M, Christ-Crain M. A Copeptin-Based Approach in the Diagnosis of Diabetes Insipidus. N Engl J Med. 2018 Aug 2;379(5):428-439. doi: 10.1056/NEJMoa1803760. PMID 30067922